CLINICAL TRIAL: NCT00174473
Title: An Open-label, Intravenous to Oral Switch, Multiple Dose Multi-Centre Study to Investigate the Pharmacokinetics, Safety and Tolerability of Voriconazole in Hospitalized Children Aged 2 to 12 Years Who Require Treatment for the Prevention of Systemic Fungal Infections.
Brief Title: A Study to Investigate the Pharmacokinetics, Safety and Tolerability of Voriconazole in Children
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A1501037
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2011-05-10 (Estimated); Status verified 2011-05

CONDITIONS: Neutropenia
MeSH Terms: conditions — Neutropenia | interventions — Voriconazole

INTERVENTIONS:
Drug: Voriconazole

SUMMARY:
This is a study to investigate the pharmacokinetics, safety and tolerability of several doses of voriconazole, intravenous and oral suspension formulations, in children

ELIGIBILITY:
Inclusion Criteria:

* Children who require a systemic antifungal agent for the prevention of systemic fungal infection

Exclusion Criteria:

* Children who are receiving medications which cannot be taken concomitantly with voriconazole.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 49 (Actual)
Dates: Start 2003-06; Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
The primary objective was to investigate the pharmacokinetics of voriconazole following intravenous (iv) to oral administration in immunocompromised children aged 2 to <12years.

SECONDARY OUTCOMES:
The secondary objective was to evaluate the safety and tolerability of multiple dose administration of voriconazole in immunocompromised children requiring treatment for the prevention of systemic fungal infection.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer